CLINICAL TRIAL: NCT01047917
Title: Meditation to Reduce Stress and Improve Quality of Life: A Feasibility Study
Brief Title: Meditation to Reduce Stress and Improve Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dietlind Wahner-Roedler, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 07-006601
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Stress
Keywords: Meditation; Relaxation Therapy; Quality of Life
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Meditation DVD (Experimental): All participants will receive a Meditation DVD to practice at home daily for a total of 4 weeks.
  Interventions: Behavioral: Meditation DVD

INTERVENTIONS:
Behavioral: Meditation DVD — Participants will undergo a one-hour group instruction session in meditation held by Dr. Amit Sood. Participants will then receive a DVD to practice the intervention at home daily for a total of 4 weeks. The DVD will have 3 different programs of 5, 15, and 30 minutes each loaded on it with a menu option to choose one of the programs.
  Other Names: Meditation

SUMMARY:
The purpose of this study is to test a simple meditation program that is easy to learn; inexpensive; easy to practice; non-religion based; and has wide applicability to multiple medical conditions. This program has been developed by the Complementary and Integrative Medicine Program at the Mayo Clinic.

DETAILED DESCRIPTION:
Stress is a ubiquitous problem and a mediator of symptoms for a variety of medical conditions. Most medical diagnoses, procedures, and physician visits are associated with considerable stress. Excessive stress is associated with adverse medical outcomes, unhealthy coping mechanisms, symptoms of anxiety and depression, and overall a poor quality of life. No specific pharmacologic treatment is available for treating stress. Further, it is often difficult or impossible to change the reality of circumstances causing stress in an individual. Thus increasing individual coping mechanisms and ability of a person to handle stress, rather than changing the stressors itself, might be a more feasible approach towards reducing stress.

Meditation is a widely used and increasingly popular intervention that positively affects the individual at cognitive, physical, emotional, behavioral, and spiritual levels. A practice of meditation has been shown to reduce symptoms of stress and improve overall quality of life. Several meditation programs exist, however most are limited by considerable expense, need for elaborate training, lack of widespread availability, or incorporation of ideas and practices unique to a particular culture.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Good general health
* Access to a DVD player
* Provided with, understand, and have signed the informed consent

Exclusion Criteria:

* Are currently using (at the time of enrollment) antipsychotics or recently (< 3 months) started on antidepressants. Patients on stable dose of antidepressant (for ≥ 3 months) will be allowed.
* Have a lifetime history of schizophrenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of incorporating a 4-week innovative meditation program into the daily activities of healthy Mayo Clinic employees for improving stress. | 4 Weeks

SECONDARY OUTCOMES:
To assess the effect of a 4-week program of meditation on perceived stress and overall quality of life compared to baseline. | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dietlind L. Wahner-Roedler, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Prasad K, Wahner-Roedler DL, Cha SS, Sood A. Effect of a single-session meditation training to reduce stress and improve quality of life among health care professionals: a "dose-ranging" feasibility study. Altern Ther Health Med. 2011 May-Jun;17(3):46-9. PMID 22164812